CLINICAL TRIAL: NCT00191022
Title: A Randomized, Double-Blind Comparison of LY686017, Paroxetine, and Placebo in the Treatment of Social Anxiety Disorder
Brief Title: Comparison of LY686017 With a Marketed Drug in the Treatment of Social Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7958; H8R-MC-HJAG
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Social Phobia
MeSH Terms: conditions — Phobia, Social | interventions — LY686017; Paroxetine

INTERVENTIONS:
Drug: LY686017
Drug: paroxetine
Drug: placebo

SUMMARY:
This study is a Phase 2 trial to test the efficacy of LY686017 in the treatment of Social Anxiety Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age and not more than 65 years of age.
* Must sign the informed consent document.
* Present at Visit 1 with social anxiety disorder based on a Clinical Global Impression-Severity score of greater than or equal to 4.
* Females of childbearing potential (not surgically sterilized and between menarche and 1 year post-menopause) must test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use both a reliable primary method of birth control.
* Judged to be reliable and willing to keep all appointments for clinic visits, tests, and procedures required by the protocol.

Exclusion Criteria:

* Have any comorbid Axis I disorders (such as major depression, obsessive compulsive disorder, post-traumatic stress disorder, or panic disorder), in the opinion of the investigator, if the disorder occurred within the last 6 months.
* Have had any previous or current diagnoses of bipolar disorders, schizophrenia, or other psychotic disorders.
* Have the presence of an Axis II disorder, except avoidant personality disorder.
* Have a serious medical illness.
* Have abnormal thyroid-stimulating hormone (TSH) concentrations or are taking thyroid supplements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185
Dates: Start 2004-12; Study Completion 2007-01

PRIMARY OUTCOMES:
Superiority is defined as a statistically greater reduction of the mean change from baseline to endpoint (after 12 weeks of treatment) in the Liebowitz Social Anxiety Scale (LSAS) total score.

SECONDARY OUTCOMES:
To compare the safety and tolerability of LY686017 with placebo during 12-week treatment.
To evaluate efficacy of LY686017 compared with placebo in treatment of social anxiety disorder during 12-week therapy based on mean improvement in the following measures:
The Liebowitz Social Anxiety subscale scores
The Clinical Global Impression-Improvement scale
The Hamilton Anxiety Scale total score and
The Clinical Global Impression-Severity scale
To assess the efficacy of LY686017 compared with placebo on health outcomes as measured by the Sheehan Disability scale.
To investigate the population pharmacokinetics of LY686017 following multiple administrations of LY686017.
To ascertain whether another approved marketed drug for
social anxiety disorder is statistically significantly more efficacious than placebo in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM to 5PM EST (UTC/GMT - 5 hours EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Burbank, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, New Britain, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Herndon, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, West Allis, Wisconsin

REFERENCES:
- [Derived] Tauscher J, Kielbasa W, Iyengar S, Vandenhende F, Peng X, Mozley D, Gehlert DR, Marek G. Development of the 2nd generation neurokinin-1 receptor antagonist LY686017 for social anxiety disorder. Eur Neuropsychopharmacol. 2010 Feb;20(2):80-7. doi: 10.1016/j.euroneuro.2009.10.005. Epub 2009 Dec 16. PMID 20018493